CLINICAL TRIAL: NCT05915871
Title: An Open-label, Fixed-sequence Study to Evaluate the Drug-drug Interactions Between Tegoprazan Tablets and Bismuth Potassium Citrate Capsules, Amoxicillin Capsules, and Clarithromycin Tablets in Healthy Subjects
Brief Title: Drug Interaction Study Between Tegoprazan, Bismuth, Amoxicillin and Clarithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NE822202
Record Dates: First submitted 2023-06-02; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan; Bismuth; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tegoprazan, Bismuth, Amoxicillin and Clarithromycin (Experimental): Oral administration of Tegoprazan 50 mg twice daily on Days 1 to 7. Oral administration of Bismuth 600 mg twice daily, Amoxicilli 1000 mg twice daily and Clarithromycin 500 mg twice daily on Days 14 to 20.
  Oral administration of Tegoprazan 50 mg twice daily, Bismuth 600 mg twice daily, Amoxicilli 1000 mg twice daily and Clarithromycin 500mg twice daily on Days 21 to 27.
  Interventions: Drug: Tegoprazan; Drug: Bismuth; Drug: Amoxicilli; Drug: Clarithromycin

INTERVENTIONS:
Drug: Tegoprazan — Tablet for oral administration
Drug: Bismuth — Capsule for oral administration
Drug: Amoxicilli — Capsule for oral administration
Drug: Clarithromycin — Tablet for oral administration

SUMMARY:
To evaluate the pharmacokinetic interaction between tegoprazan and combination of Amoxicillin, Clarithromycin and bismuth in healthy adult volunteers.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic interaction between tegoprazan and combination of Amoxicillin, Clarithromycin and bismuth in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects fully understand the objectives, nature, method, possible AEs of the trial, voluntarily participate in this clinical study, sign the ICF in person prior to the start of any study procedure, and promise that they will participate in all the study procedures in person.

  2. Chinese healthy male and non-lactating female subjects who are 18 to 55 years of age (inclusive) at the signing of ICF.

  3. Body mass index (BMI) of 19.0 to 28.0 kg/m2 (inclusive); and male weight ≥ 50.0 kg, female weight ≥ 45.0 kg.

  4. Subjects can communicate well with the investigator and understand and comply with various requirements of the study.

Exclusion Criteria:

* 1. Diseases with prior and current abnormal clinical manifestations to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, and bones.

  2. People with a history of specific allergy (asthma, urticaria, eczema, etc.), an allergic constitution, or known hypersensitivity to tegoprazan, bismuth potassium citrate, amoxicillin, clarithromycin, penicillin, and macrolide antibiotics, or hypersensitivity to any ingredient of the drug products.

  3. Positive reaction to penicillin skin test. 4. History of active ulcer or significant hemorrhage from gastrointestinal tract, genitourinary tract or respiratory tract, or central nervous system hemorrhage.

  5. History of dysphagia or any gastrointestinal disorder affecting drug absorption (as judged by the investigator).

  6. Surgery within 3 months prior to screening, or planning to receive surgery during the study, and history of any surgery that may affect drug absorption (e.g., gastrectomy).

  7. Intolerance to venipuncture, or history of fear of needles or blood. 8. Lactose intolerance (history of diarrhea due to drinking milk). 9. History of illicit drug abuse within 6 months prior to screening, history of illicit drug use, or urine drug screen test positive.

  10. Mean alcohol use > 14 units of alcohol (1 unit of alcohol ≈ 360 mL of beer, 150 mL of wine, or 45 mL of spirit) per week within 3 months prior to screening, or alcohol breath test positive, or inability to stop drinking during the trial period.

  11. Mean daily smoking > 5 cigarettes within 3 months prior to screening, or inability to stop using any tobacco products during the trial period.

  12. Participation in any clinical trial of other investigational drug/device within 3 months prior to the first dose of study drug, or participation in 3 or more drug/device clinical trials in the past one year; if the half-life of other study drugs is long (5 half-lives exceed 3 months), the time interval required will be longer, i.e., 5 half-lives of the drug.

  13. Blood donation including donating blood components or massive blood loss (≥ 200 mL) within 3 months prior to screening; blood transfusion or use of blood products within 3 months prior to screening.

  14. History of vaccination within 1 month prior to screening, or planned vaccination during the study period.

  15. Use of any drugs inhibiting or inducing hepatic drug metabolism within 28 days prior to first dose of study drug.

  16. Use of any prescription drugs, over-the-counter drugs, dietary supplements, or Chinese herbal medicines within 14 days prior to first dose.

  17. Any of the hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody, or anti-Treponema pallidum specific antibody tests is positive.

  18. At the time of screening, the results of vital signs (blood pressure, pulse rate, and body temperature), physical examination, and laboratory tests (complete blood count, blood chemistry, coagulation, and urinalysis) are judged as abnormal and clinically significant by the investigator.

  19. In the supine 12-lead ECG performed after at least 10 minutes of quiet rest during screening, QT interval corrected by Fridericia's formula (QTcF) > 470 msec (female)/450 msec (male) [Fridericia's formula is QTcF = QT/(RR)1/3] or QRS complex > 120 msec [if the QTcF of the 1st measurement exceeds 450 msec (female QTcF > 470 msec) or QRS > 120 msec, 12-lead ECG measurements should be repeated 2 times, and a judgment should be made using the mean QTcF or QRS value of the 3 measurements].

  20. Subjects with a history of prolonged QT interval or ventricular arrhythmia (including torsade de pointes).

  21. Subjects with hypokalemia (at risk of prolonged QT interval). 22. Creatinine clearance (CLCr) < 90 mL/min. The calculation method of creatinine clearance is shown in Appendix 4.

  23. Subjects who cannot stop taking strenuous exercise within 48 hours prior to first dose of study drug and during the trial period.

  24. Subjects who consume any alcohol-containing, caffeine-containing, or xanthine-rich food or beverage within 48 hours prior to first dose of study drug; or cannot stop consuming such products during the trial period.

  25. Subjects who consume pitaya, mango, grapefruit, or grapefruit-related citrus fruits (e.g., pomegranate, starfruit, Seville orange, and pomelo) or food or beverage prepared from such fruits within 7 days prior to first dose of study drug, or cannot stop taking these fruits or food or beverage prepared from them during the trial period.

  26. Subject or his/her partner has planned parenthood, or is unwilling to take effective contraceptive measures (see Appendix 1 for details), or has a sperm or egg donation plan throughout the study and within 3 months after last dose of study drug. Female subjects who do not take effective contraceptive measures within 15 days prior to screening.

  27. Female subjects who have a positive blood pregnancy test at screening. 28. Unwillingness or inability to follow the lifestyle guidance (e.g., dietary restrictions and activity requirements) described in the study protocol.

  29. Subjects have other acute or chronic medical or psychiatric disorders and thereby are judged by the investigator as not suitable for participating in this study, which may increase the risk related to this study or may interfere with the interpretation of study results.

  30. Other subjects who are judged unsuitable for participation in the clinical trial by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
AUCtau of Tegoprazan, Bismuth, Amoxicillin, and Clarithromycin Following Multiple Oral Doses | Up to Day 27
  Area under the curve over a 12-hour dosing interval at steady state (AUCtau)
Cmax,ss of Tegoprazan, Bismuth, Amoxicillin, and Clarithromycin Following Multiple Oral Doses | Up to Day 27
  Steady state maximum concentration (Cmax,ss)

SECONDARY OUTCOMES:
Tmax,ss of tegoprazan, bismuth, amoxicillin, and clarithromycin | Up to Day 27
  steady-state time to reach maximum concentration (Tmax,ss)
T1/2 of tegoprazan, bismuth, amoxicillin, and clarithromycin | Up to Day 27
  elimination half-life (t1/2)
CL/F of tegoprazan, bismuth, amoxicillin, and clarithromycin | Up to Day 27
  apparent clearance (CL/F)
Vdss/F of tegoprazan, bismuth, amoxicillin, and clarithromycin | Up to Day 27
  apparent volume of distribution (Vdss/F)
Cmax,ss of M1 (tegoprazan metabolite) and 14-hydroxyclarithromycin | Up to Day 27
  Steady state maximum concentration (Cmax,ss)
AUCtau of M1 (tegoprazan metabolite) and 14-hydroxyclarithromycin | Up to Day 27
  Area under the curve over a 12-hour dosing interval at steady state (AUCtau)
Tmax,ss of M1 (tegoprazan metabolite) and 14-hydroxyclarithromycin | Up to Day 27
  steady-state time to reach maximum concentration (Tmax,ss)
T1/2 of M1 (tegoprazan metabolite) and 14-hydroxyclarithromycin | Up to Day 27
  elimination half-life (t1/2)
Number of Participants With Adverse Events | Up to Day 34
Number of Participants With Clinically Notable Electrocardiogram (ECG) Values | Up to Day 28
Number of Participants With Clinically Notable Laboratory Tests | Up to Day 28
Number of Participants With Clinically Notable Vital Signs | Up to Day 28
Number of Participants With Clinically Notable Physical Exam | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China